CLINICAL TRIAL: NCT02656927
Title: Evaluation of a Specialized Yoga Program for Persons With Spinal Cord Injury: A Randomized Controlled Trial
Brief Title: Evaluation of a Specialized Yoga Program for Persons With Spinal Cord Injury (SCI)
Acronym: SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sander Hitzig, Affiliate Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UHN-REB#15-9413-D
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Yoga; Psychological Flexibility; Mindfulness; Pain
MeSH Terms: conditions — Spinal Cord Injuries; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Condition (Experimental)
  Interventions: Behavioral: Yoga Condition
- Wait-list Control Condition (Placebo Comparator)
  Interventions: Behavioral: Yoga Condition

INTERVENTIONS:
Behavioral: Yoga Condition

SUMMARY:
The purpose of this randomized controlled study is to evaluate psychological variables, mindfulness, and pain in the context of a specialized yoga program for individuals with SCI. Participants will be randomized to either a wait-list control condition or to a specialized yoga program condition.

ELIGIBILITY:
Inclusion Criteria:

1. have an SCI or a spinal related condition,
2. be 18 years of age or older,
3. be able to speak and read English,
4. commit to two weekly, one hour yoga classes for six weeks,
5. be referred from a clinician on the inter-disciplinary team,
6. have a sitting tolerance of one hour,
7. be able to participate in gentle physical activity in that time,
8. be aware of and understand his/her health contraindications (is able to practice safely),
9. provide a note from their physician indicating that it is safe for them to participate in a physical activity intervention, such as yoga.

Exclusion Criteria:

1. are not medically stable,
2. have pre-existing medical contraindications,
3. have cognitive limitations or language comprehension issues that would impact participation (determined by care team),
4. have had a regular yoga practice in the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire-II (AAQ-II) | Change from Baseline, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change from Baseline, 6 weeks, 12 weeks
General Self-Efficacy Scale (GSES) | Change from Baseline, 6 weeks, 12 weeks
Post-Traumatic Growth Inventory-SF (PTGI-SF) | Change from Baseline, 6 weeks, 12 weeks
Connor-Davidson Resilience Scale-10 Item (CS-RISC-10) | Change from Baseline, 6 weeks, 12 weeks
Five Facet Mindfulness Questionnaire-SF (FFMQ-SF) | Change from Baseline, 6 weeks, 12 weeks
Self-Compassion Scale-SF (SCS-SF) | Change from Baseline, 6 weeks, 12 weeks
Brief Pain Inventory-SF (BPI-SF) | Change from Baseline, 6 weeks, 12 weeks
Pain Catastrophizing Scale (PCS) | Change from Baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sander L. Hitzig, PhD, Principal Investigator — University Health Network, University of Toronto; Kathryn J. Curtis, MA, Study Director — York University

IPD SHARING:
Plan to Share IPD: No